CLINICAL TRIAL: NCT01790854
Title: Bless Study (BLeeding Events and Maintenance DoSe of PraSugrel)
Brief Title: BLeeding Events and Maintenance DoSe of PraSugrel
Acronym: BLESS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low events rate. Scarce economical resources
Sponsor: David Antoniucci (Other)
Collaborators: A.R. CARD Onlus Foundation (Other)
Responsible Party: Sponsor-Investigator, David Antoniucci, Head Division of Invasive Cardiology, Careggi Hospital
Organization: Careggi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLESS Study
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Adverse Reaction to Antiplatelet Agent; Acute Coronary Syndrome
Keywords: prasugrel; antiplatelet; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel dose 5 mg/day (Experimental): 225 patients will be treated with 325 mg of aspirin (followed by a maintenance dosage of 100 mg of aspirin for at least 1 year and with 60 mg loading dose of prasugrel followed by a maintenance dosage of 5 mg/day of prasugrel for 12 months
  Interventions: Drug: Prasugrel dose 5 mg/day
- Prasugrel dose 10 mg/day (Active Comparator): 225 patients will be treated with 325 mg of aspirin (followed by a maintenance dosage of 100 mg of aspirin for at least 1 year and with 60 mg loading dose of prasugrel followed by a maintenance dosage of 10 mg/day of prasugrel for 12 months
  Interventions: Drug: Prasugrel dose 10 mg/day

INTERVENTIONS:
Drug: Prasugrel dose 5 mg/day
  Arms: Prasugrel dose 5 mg/day
Drug: Prasugrel dose 10 mg/day
  Arms: Prasugrel dose 10 mg/day

SUMMARY:
Aim: to verify if after the acute phase of ACS acute coronary syndrome (1-months), from 1 to 12 months the reduction of maintenance dose of prasugrel from 10 mg to 5 mg/day may reduce the bleeding events (5 mg vs 10 mg). All patients will be treated with 325 mg of aspirin followed by a maintenance dosage of 100 mg of aspirin for at least 1 year. At baseline (after 60 mg loading dose of prasugrel) and after 1 month (7 days after the randomization at 10 or 5 mg of prasugrel) all patients will undergo light transmittance aggregometry (LTA) test to evaluate residual platelet reactivity (pharmacodynamic effects).

ELIGIBILITY:
Inclusion Criteria:

* all ACS patients treated with PCI (percutaneous coronary intervention) and dual antiplatelet therapy (DAPT: aspirin plus prasugrel).
* Informed written consent

Exclusion Criteria:

* Age < 18 years
* Active bleeding; bleeding diathesis; coagulopathy
* History of gastrointestinal or genitourinary bleeding <2 months
* Major surgery in the last 6 weeks
* History of intracranial bleeding or structural abnormalities
* Suspected aortic dissection
* Any previous TIA (transient ischemic attack)/stroke
* Administration in the week before the index event of clopidogrel, ticlopidine, prasugrel, ticagrelor, thrombolytics, bivalirudin, low-molecular weight heparin or fondaparinux .
* Known relevant hematological deviations: Hb <10 g/dl, Thrombocytopenia. <100x10^9/l
* Use of coumadin derivatives within the last 7 days
* Chronic therapy with prasugrel or ticagrelor
* Known malignancies or other comorbid conditions with life expectancy <1 year
* Known severe liver disease, severe renal failure
* Known allergy to the study medications
* Pregnancy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
bleeding | 12 months
  major, minor and minimal bleeding defined according BARC (Bleeding Academic Research Consortium criteria (11), occurring from 1 month to the end of the study.

SECONDARY OUTCOMES:
MACE | 12 months
  MACE (cardiac death, Myocardial Infarction, stroke) occurring from 1 month to the end of the study; late stent thrombosis.

OTHER OUTCOMES:
pharmacodynamic effects | 12 months
  pharmacodynamic effects of shifting prasugrel maintenance dose from 10 mg to 5 mg after ACS
residual platelet reactivity (LTA) | baseline - 1 month
  correlation between residual platelet reactivity (LTA), both at baseline and at 1-month, with bleeding and ischemic events

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Principal Investigator — Careggi Hospital, division of Invasive Cardiology
Locations (1):
- Careggi Hospital, Florence, Italy

REFERENCES:
- [Derived] Carrabba N, Parodi G, Marcucci R, Valenti R, Gori AM, Migliorini A, Comito V, Bellandi B, Abbate R, Gensini GF, Antoniucci D. Bleeding events and maintenance dose of prasugrel: BLESS pilot study. Open Heart. 2016 Oct 31;3(2):e000460. doi: 10.1136/openhrt-2016-000460. eCollection 2016. PMID 27843564